CLINICAL TRIAL: NCT07228689
Title: Artificial Intelligence for Onsite Cytology Evaluation in Endoscopic Ultrasound
Brief Title: AI for Onsite Cytology Evaluation in Endoscopic Ultrasound
Status: Recruiting | Type: Observational
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 2343877
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Gastrointestinal Neoplasm; Mass Lesion
Keywords: endoscopic ultrasound; solid mass lesion; artificial intelligence; fine needle biopsy
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interpretation of cytology specimen by cytopathologist onsite: The interpretation of the cytology specimens will be made onsite by the cytopathologist
  Interventions: Diagnostic Test: EUS-guided fine needle biopsy
- Interpretation of cytology specimen by artificial intelligence: The interpretation of the cytology specimens will be made onsite by the AI program
  Interventions: Diagnostic Test: EUS-guided fine needle biopsy

INTERVENTIONS:
Diagnostic Test: EUS-guided fine needle biopsy — EUS-guided fine needle biopsy of solid mass lesions in the gastrointestinal tract

SUMMARY:
The aim of this study is to determine if the widely available artificial intelligence platform ChatGPT can accurately identify the abnormalities present on cytology specimens obtained at EUS-FNB of solid mass lesions in the gastrointestinal tract, in comparison with interpretation by cytopathologists as the gold standard.

DETAILED DESCRIPTION:
The diagnostic accuracy of EUS-guided fine needle biopsy of lesions in the gastrointestinal tract is dependent on the availability of a cytopathologist to render a rapid on-site evaluation (ROSE), with studies showing that the presence of an on-site cytopathologist improves the diagnostic yield, decreases the number of inadequate or unsatisfactory samples, and limits the number of passes required to establish a diagnosis. However, the availability of ROSE is variable across centers and regions, with the availability of onsite cytopathology services limited to a handful of tertiary referral centers in the United States.

ChatGPT is a universally available, generative artificial intelligence program developed by OpenAI. The aim of this study is to determine if this AI platform can accurately identify the abnormalities present on cytology specimens obtained at EUS-FNB of solid mass lesions in the gastrointestinal tract, in comparison with interpretation by cytopathologists as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or greater
* Patients undergoing EUS-guided fine needle biopsy of solid mass lesions in the gastrointestinal tract

Exclusion Criteria:

* Age less than 18 years
* Patients not undergoing sampling of solid mass lesions at EUS
* Patients with cystic lesions in the gastrointestinal tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or greater, undergoing EUS-guided fine needle biopsy of solid mass lesions in the gastrointestinal tract.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy at rapid onsite evaluation | 1 day
  The ability of the AI system to correctly interpret cytology images, compared to cytopathologists.

SECONDARY OUTCOMES:
Diagnostic accuracy compared to final pathology | 7 days
  The ability of the AI system to corrently interpret cytology images, compared to final pathology results.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Bang, MD MPH, Principal Investigator — Orlando Health
Locations (1):
- Orlando Health Digestive Health Institute, Orlando, Florida, United States